CLINICAL TRIAL: NCT05957796
Title: The Utility of a Novel Eye Shield With Reusable Adhesive Anchors for Post-operative Care After Ophthalmic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Augusta University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2024576
Record Dates: First submitted 2023-06-16; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Cataract; Eye Disease
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Regular eye shield after surgery (Active Comparator): Alcon eye shield after surgery
  Interventions: Other: Standard Alcon Eye Shield
- Novel prototype eye shield after surgery (Experimental): Novel prototype eye shield after surgery
  Interventions: Device: Novel "Snaps" Eye Shield

INTERVENTIONS:
Device: Novel "Snaps" Eye Shield — Using a novel eye shield, "Snaps" manufactured in Morgantown, WV by Intermed Labs after cataract surgery that has a different adhesive mechanism that utilizes adhesive and snap-on attachments to the shield.
  Arms: Novel prototype eye shield after surgery
Other: Standard Alcon Eye Shield — Use normal Alcon eye shield with tape to adhere to shield to eye postop.
  Arms: Regular eye shield after surgery

SUMMARY:
The purpose of this research study is to evaluate the efficacy, patient preference, and utility of a novel eye shield that utilizes a different adhesive mechanism in comparison to the current standard of care. The aims are to see if this product could be incorporated into postoperative care in the future to improve patient satisfaction and compliance.

The study will involve 20 patients during the postoperative timeframe after cataract extraction and intraocular lens placement (CEIOL). These patients will be chosen from the clinic of Dr. Marc Toeteberg who will plan to have both eye surgeries done within 3 months of each other. These patients will be randomized to either control or intervention group. Intervention group will receive our novel eye shield prototype, while control group will receive an Alcon plastic eye shield. Both groups will receive the eye shields after surgery and will be sent home with these eye shields with normal postoperative care directions. Patient will be directed to wear eye shields for 24 hours then at night for first 2 weeks after surgery, while adhering to postoperative eye drops regimen.

After successfully healing and passing the postoperative timeframe for the first eye we will proceed to the second arm of the study. Approximately 1-2 months after healing from the first surgery, patient will be scheduled for cataract surgery on the other eye, as is standard of care. After surgery on the second eye the patient will be given the other eye shield than what they received after the first surgery (control groups will receive the novel eye shield and experimental groups will receive the control eye shield). They will proceed to follow identical postoperative protocols after the second surgery. A short quantitative and qualitative questionnaire directly comparing the two eye shield experiences will be provided at the 1 month follow-up after the eye surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female cataract surgery patients of 18 years or older, with surgical plans for cataract extraction via phacoemulsification and intraocular lens placement. Patient must be having plans to have both eye cataracts removed surgically in succession within 3 months of each other.

Exclusion Criteria:

* Patients receiving more advanced intraocular surgery, even if that surgery includes cataract removal and intraocular lens placement, including trabeculectomy, microinvasive glaucoma surgery, vitrectomy, or any other ophthalmic procedure. Pregnancy also an exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of use of a new eye shield versus regular eye shield. | Over the course of the 2 cataract surgeries, approximately taking 3 months including preoperative and postoperative care.
  This primarily focuses on comfort and satisfaction to the patient between the two shields. This will be assessed via a questionnaire using a likert scale to get quantitative data from the questions.

CONTACTS AND LOCATIONS:
Locations (1):
- Augusta University, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No